CLINICAL TRIAL: NCT04206748
Title: iGlucose® Remote Patient Monitoring Device as an Adjunct to Routine Glucose Meter Devices for Glycemic Management and Control in Gestational Diabetes: a Pilot Randomized, Controlled Trial
Brief Title: iGlucose® Remote Patient Monitoring Device as an Adjunct to Routine Glucose Meter Devices for Glycemic Management and Control in Gestational Diabetes
Acronym: iGlucose
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Smart Meter Corporation (Industry)
Responsible Party: Principal Investigator, Joycelyn Ashby Cornthwaite, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MS-19-0402
Record Dates: First submitted 2019-11-15; First posted 2019-12-20 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Gestational Diabetes; Type2 Diabetes; Pregnancy in Diabetic
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy in Diabetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- iGlucose Smart Meter (Experimental)
  Interventions: Device: iGlucose Smart Meter System
- Rx glucose meter (Placebo Comparator)
  Interventions: Device: Routine Care-RX meter

INTERVENTIONS:
Device: iGlucose Smart Meter System — Subjects will have routine care enhanced by use of theThe iGlucose Smart meter system. This is an example of integration of a SMBG system with internet-based technology; including cell phone notifications for reminders, feedback, and communication with clinicians
  Arms: iGlucose Smart Meter
Device: Routine Care-RX meter — Subjects will receive routine care with the insurance prescribed glucose meter. They will self manage with traditional diabetes diary.
  Arms: Rx glucose meter

SUMMARY:
The purpose of this study is to investigate whether automation of glucose monitoring data to facilitate the total number of recommended and completed SMBG checks improve clinical outcomes for women living with gestational and type 2 diabetes during pregnancy? This is a RCT

ELIGIBILITY:
Inclusion Criteria

* All patients >/= women 18 years of age with gestational diabetes or type 2 diabetes during pregnancy and identified by the research team and consented before 30.6 weeks.
* Non-anomalous singletons
* Ability to provide informed consent

Exclusion Criteria

* Patients with Type 1 diabetes
* Patients with fetal major congenital abnormalities
* Patients identified/referred after 30.6 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-11-12 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Neonatal morbidity | at the time of discharge (about 2-7 days after birth)
Neonatal gestational age at delivery | at delivery
# of neonates who where Small for gestational age (SGA) | at delivery
Neonatal intensive care unit (NICU) length of stay | delivery to discharge (2-7 days)
# of Neonates with hyperbilirubinemia-requiring therapy. | delivery to discharge (2-7 days)

SECONDARY OUTCOMES:
Average Neonatal Weight | at the time of discharge (about 2-7 days after birth)
  To evaluate the relationship of change in average neonatal weight to two skill sets of Self-monitoring of blood glucose (SMBG), operational and interpretive, as demonstrated by patient-perceived self-efficacy and adherence to self-care behaviors
Maternal Mean fasting glucose | perinatal to postpartum (32 weeks)
Maternal Mean post prandial glucose | perinatal to postpartum (32 weeks)
Maternal # of Hypoglycemia events (<60 mg/dl) | perinatal to postpartum (32 weeks)
Maternal weight gain during pregnancy | perinatal to postpartum (32 weeks)
Maternal Gestational hypertension | perinatal to postpartum (32 weeks)
Maternal Preeclampsia | perinatal to postpartum (32 weeks)
Maternal Cesarean delivery | at delivery
Maternal Operative vaginal delivery | at delivery
Effect of SMBG checks on pregnancy | perinatal to postpartum (32 weeks)
  To evaluate relationship between percent of total achieved SMBG checks, diabetes distress, and maternal and neonatal outcomes, for women living with GDM and T2DM during pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No